CLINICAL TRIAL: NCT01953575
Title: Mucosal Impedance in Eosinophilic Esophagitis and the Effect of Treatment
Brief Title: Mucosal Impedance and Eosinophilic Esophagitis
Acronym: EoE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, David A. Katzka, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 13-005778
Record Dates: First submitted 2013-09-26; First posted 2013-10-01 (Estimated); Results first posted 2020-04-15 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Eosinophilic Esophagitis
Keywords: Mucosal Impedance; Eosinophilic Esophagitis; EoE
MeSH Terms: conditions — Eosinophilic Esophagitis | interventions — Gastroscopy; Endoscopy, Digestive System

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Active Eosinophilic Esophagitis (Experimental): Subjects with an eosinophil count greater than 15 eosinophil per high-powered field (Eos/HPF) and do not have trouble swallowing during the clinical endoscopy
  Interventions: Device: Mucosal Impedance; Procedure: Upper Endoscopy
- Inactive Eosinophilic Esophagitis (Experimental): Subjects with an eosinophil count less than 15 eosinophil per high-powered field (Eos/HPF) and do not have trouble swallowing during the clinical endoscopy
  Interventions: Device: Mucosal Impedance; Procedure: Upper Endoscopy
- Control group (Placebo Comparator): Subjects are those undergoing clinically indicated upper endoscopy for nonesophageal symptoms in whom a normal-appearing esophagus was found at the time of endoscopy
  Interventions: Procedure: Upper Endoscopy

INTERVENTIONS:
Device: Mucosal Impedance — A tiny tube will be placed through the endoscope into the esophagus. 5 cm above where the stomach and esophagus meet for 5 seconds. At 10 cm above where the stomach and esophagus meet the catheter will be placed for 5 seconds. And at 20 cm above where the stomach and esophagus meet the catheter will be placed for 5 seconds.
  Other Names: ph impedance; ph monitor
  Arms: Active Eosinophilic Esophagitis; Inactive Eosinophilic Esophagitis
Procedure: Upper Endoscopy — Esophagogastroduodenoscopy, also called by various other names, is a diagnostic endoscopic procedure that visualizes the upper part of the gastrointestinal tract down to the duodenum.
  Other Names: Esophagogastroduodenoscopy (EGD)

SUMMARY:
Do patients with eosinophilic esophagitis have baseline increased esophageal mucosal impedance?

And will treatment that reverses esophageal eosinophilia in patients, correct abnormalities in mucosal impedance?

ELIGIBILITY:
Inclusion criteria:

* Adults ages 18-90 undergoing clinically indicated upper endoscopy
* Patients with EoE, defined as dysphagia with histologic finding of greater than or equal to 15 eosinophils per high powered field on esophageal biopsy despite at least 6 weeks of twice daily proton pump inhibitor therapy
* Patients undergoing clinically indicated upper endoscopy for indications other than dysphagia or Gastroesophageal reflux disease (GERD) with normal appearing esophageal mucosa.

Exclusion criteria:

* Medical conditions such as severe heart or lung disease that preclude safe performance of endoscopy
* Patients with conditions known to be associated with esophageal eosinophilia, including Crohn's disease, Churg-Strauss, achalasia, and hypereosinophilic syndrome
* Inability to read due to: Blindness, cognitive dysfunction, or English language illiteracy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-09; Primary Completion 2019-06-10 (Actual); Study Completion 2019-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Katzka, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Eosinophilic Esophagitis | Inactive Eosinophilic Esophagitis | Control Group
Started | 10 | 10 | 10
Completed | 10 | 10 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Eosinophilic Esophagitis | Inactive Eosinophilic Esophagitis | Control Group | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Continuous [Median (Full Range); unit: years] | 41 [24 to 62] | 46 [18 to 64] | 37 [19 to 52] | 41 [18 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 6 | 10
  Male | 8 | 8 | 4 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 10 | 10 | 10 | 30
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 10 | 30

OUTCOME MEASURES:

1. Primary Outcome: Esophageal Mucosal Impedance (MI)
Description: An endoscopically placed probe measured electrical impedance of the esophageal lining by direct mucosal contact. Impedance measurements of the esophageal mucosa were expressed in ohms as the ratio of voltage to current Impedance measurements were obtained at 2, 5, 10, and 15 cm above the gastroesophageal junction.
Time Frame: baseline to one year
Measure: Mean (Inter-Quartile Range); unit: Ohms
Arm/Group | Active Eosinophilic Esophagitis | Inactive Eosinophilic Esophagitis | Control Group
Number analyzed (Participants) | 10 | 10 | 10
Ohms
  2cm | 1457 [973 to 1794] | 3463 [2313 to 3980] | 4225 [3546 to 6733]
  5cm | 1713 [1243 to 2702] | 5110 [3968 to 6406] | 4741 [3575 to 7613]
  10cm | 1731 [1131 to 2180] | 4500 [3500 to 6400] | 5943 [4581 to 7843]
  15cm | 1791 [1244 to 4602] | 3378 [2243 to 5125] | 6033 [3742 to 6841]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline endoscopy to end of study, for a total of approximately 1 year.
Arm/Group | Active Eosinophilic Esophagitis | Inactive Eosinophilic Esophagitis | Control Group
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-02-02): https://cdn.clinicaltrials.gov/large-docs/75/NCT01953575/Prot_SAP_000.pdf